CLINICAL TRIAL: NCT06643975
Title: Assessment of Patient Satisfaction and Crestal Bone Changes Around One-piece Zirconia and Titanium Implants in Mandibular Implant-Retained Overdenture: A Randomized Clinical Trial
Brief Title: Patient Satisfaction and Crestal Bone Changes Around One-piece Zirconia(Zr) and Titanium(Ti) in Implant-Retained Mandibular Overdenture
Acronym: (Zr) - (Ti)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammad Eissa Mohammad Irakky, Assistant Lecturer of oral and maxillofacial prosthodontics, faculty of dentistry , Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1372
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Complete Edentulism
Keywords: Zirconia; One-piece; Overdenture; Implant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium dental implants group (Active Comparator): Two-implants One-piece titanium dental implants with titanium ball attachments retaining mandibular overdentures
  Interventions: Other: One-piece titanium dental implants
- Zirconia dental implants group (Active Comparator): Two-implants One-piece zirconia dental implants with zirconia ball attachments retaining mandibular overdentures
  Interventions: Other: One-piece zirconia dental implants

INTERVENTIONS:
Other: One-piece zirconia dental implants — One-piece zirconia dental implants with zirconia ball attachments, these implants are metal free made of oxide ceramics with cutting-edge Selective laser melting(SLM) surface treatment technology
  Other Names: Z-SYSTEMS; ceramic implants
  Arms: Zirconia dental implants group
Other: One-piece titanium dental implants — One-piece Titanium dental implants with titanium ball attachments, these implants are gold standard compatible implants
  Arms: Titanium dental implants group

SUMMARY:
This interventional randomized clinical trial study is conducted to assess patient satisfaction and crestal bone changes around one-piece Zr and Ti Implants in mandibular implant-retained overdenture in completely edentulous male patients in the age group between (50-60)years old to know if there will be a significant difference between the two types of dental implants through 12 months after the definitive prosthetic loading

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* The age range of 50 to 60 years old (average of 55).
* moderately developed mandibular residual ridges, covered with healthy mucosa, firmly attached to the underling bone and with average mucosal thickness (2-3) mm.
* At least 12 mm of vertical bone height in the mandible allowing for placement of a 10 mm implant (2 mm safety distance to inferior alveolar nerve).
* Patients were selected with Angle class-I maxillomandibular relationship with sufficient inter-arch space (13-15mm

Exclusion Criteria:

* Heavy smokers of more than 10 cigarettes a day
* Poor oral hygiene.
* Patients with temporomandibular joint disorders(TMD),
* Patients suffered of xerostomia,
* Patients exhibited Para-functional habits, or recent extractions were excluded.
* Patients with systemic diseases that might affect bone quality or quantity, or retard healing of the surgical wounds were excluded.
* Patients receiving intravenous forms of bisphosphonates.
* Patients who have had radiation therapy to the head and neck region.
* Patients with existing implants in the jaws
* Patients with previous bone grafting in either the maxillary or mandibular jaws.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Crestal bone changes | 12 months
  Measuring the amount of marginal(crestal) bone changes either loss or gain around the dental implants using the cone beam computed tomography(CBCT) in millimeter scales about the original marginal bone height measured at the time of the visit of final (definitive) prosthetic loading.
  The positive(+ve) values mean an increase (gain) in the marginal bone height around the implants, the more the +ve value, the more the gain in the bone height which is the better outcome, while the negative (-ve) values mean decrease (loss) in the marginal bone height around the implants, the more the -ve value, the more loss in the bone height, which is the worse outcome.

SECONDARY OUTCOMES:
Patients Satisfaction | 12 months
  measuring the degree of patient satisfaction using a Patient's Denture Assessment (PDA) questionnaire, via a Likert scale which uses a 5-point system from 1 to 5, All items are scored as follows: unsatisfactory =1 hardly satisfactory =2 moderately satisfactory=3 very satisfactory=4 excellent satisfaction=5 The greater (higher) the score, the more patient satisfaction, which is the better outcome, while the weaker (lower) the score, the less is patient satisfaction, which is the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Irakky, masters, Principal Investigator — Faculty of Dentistry, Benha University; Omnia M. Refai, PHD, Study Director — Faculty of Dentistry, Ain Shams Univeristy; Noha Helmy Nawar, PHD, Study Director — Faculty of Dentistry, Ain Shams Univeristy
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt